CLINICAL TRIAL: NCT07207070
Title: A Randomised, Open-label, Multicentre Phase III Clinical Study to Evaluate the Efficacy and Safety of JS105 Combined With Dalpiciclib and Fulvestrant Compared With Dalpiciclib and Fulvestrant in Patients With PIK3CA-mutated, HR-positive, HER2-negative Recurrent or Metastatic Breast Cancer.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Risen (Suzhou) Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS105-004-III-BC
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib; Fulvestrant

STUDY DESIGN:
Intervention Model Description: Experimental group：JS105:Dose according to the protocal, orally, once daily (QD), administered continuously. Dalpiciclib :Dose according to the protocal, orally, QD, taken for 3 weeks, followedby 1 week off in each 4-week cycle； Fulvestrant Dose according to the protocal, administered intramuscularly on day 1 and day 15 of the first cycle and then on day 1 of each subsequent 4-week cycle.
  Control group：Dalpiciclib : Dose according to the protocal, orally, QD, taken for 3 weeks, followed by 1 week off in each 4-week cycle；Fulvestrant: Dose according to the protocal, administered intramuscularly on day 1 and day 15 of the first cycle and then on day 1 of each subsequent 4-week cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS105+Dalpiciclib+Fulvestrant (Experimental): Patients will receive JS105, Dalpiciclib and Fulvestrant.
  Interventions: Drug: JS105; Drug: Dalpiciclib; Drug: Fulvestrant 50 Mg/mL Intramuscular Solution
- Dalpiciclib+Fulvestrant (Active Comparator): Patients will receive Dalpiciclib and Fulvestrant.
  Interventions: Drug: Dalpiciclib; Drug: Fulvestrant 50 Mg/mL Intramuscular Solution

INTERVENTIONS:
Drug: JS105 — Patients will receive oral JS105 on Days 1-28 of each 4-week cycle.
  Arms: JS105+Dalpiciclib+Fulvestrant
Drug: Dalpiciclib — Patients will receive oral Dalpiciclib for 3 weeks, followed by 1 week off in each 4-week cycle；
Drug: Fulvestrant 50 Mg/mL Intramuscular Solution — Patients will receive intramuscular Fulvestrant on day 1 and day 15 of the first cycle and then on day 1 of each subsequent 4-week cycle.

SUMMARY:
This study is a randomised, open-label, multicentre phase III clinical study evaluating the efficacy and safety of JS105 combined with Dalpiciclib and Fulvestrant compared with Dalpiciclib and Fulvestrant in patients with PIK3CA-mutated, HR-positive, HER2-negative recurrent or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the consent form, age must be between 18 and 75 years old, males and females;
2. Patients with unresectable PIK3CA-mutated HR-positive HER2-negative recurrent or metastatic breast cancer;
3. Consent to provide tumour tissue or blood samples to determine the PIK3CA mutation status;
4. ECOG 0 or 1;
5. At least one measurable lesion as per RECIST v1.1, or only bone metastases;
6. Expected survival≥12 weeks;
7. Good organ function;
8. Patients voluntarily join the study and sign the informed consent;

Exclusion Criteria:

1. Previously treated with fulvestrant or PI3K/AKT/mTOR inhibitors;
2. Presence of untreated or active central nervous system (CNS) metastases;
3. Presence of significant clinical symptoms or uncontrolled pleural effusion, ascites, or pericardial effusion that require repeated drainage (once a month or more frequently);
4. Untreated spinal cord compression, or previously treated spinal cord compression without clinical evidence of disease stability for at least 4 weeks prior to the first study treatment;
5. Have received other anti-tumor treatment within 2-4 weeks before the first dose;
6. Toxicities from prior anti-tumor therapy that have not recovered to ≤ Grade 1;
7. Coexisting uncontrolled accompanying diseases, including but not limited to: history of type I diabetes or uncontrolled type II diabetes, presence of active infection, severe cardiovascular or cerebrovascular diseases, etc;
8. Having another malignant tumour within the last 5 years prior to the first study treatment, except for malignancies that are expected to be cured after treatment;
9. Active hepatitis B or C;
10. Known hypersensitivity to any of the study drugs or their excipients;
11. Pregnant or breastfeeding females;
12. Presence of other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participation in the study, affect treatment compliance, or interfere with study results, as judged by the investigator;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Blind Independent Central Review (BICR) assessed PFS based on RECIST v1.1 (BICR-PFS) | Up to 3.5 years
  PFS is defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first).

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years
  OS is defined as the time from randomization to death from any cause.
Investigator-assessed Progression-Free Survival (PFS) | Up to 3.5 years
  PFS is defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first).
1-year and 2-year Progression-Free Survival (PFS) rate | Up to 3.5 years
  1-year and 2-year Progression-Free Survival (PFS) rate
Objective Response Rate (ORR) | Up to 5 years
  Objective Response Rate (ORR) as Assessed by Investigator or BICR according to RECIST v1.1
Duration of Objective Response (DOR) | Up to 5 years
  Duration of Objective Response (DOR) as Assessed by Investigator or BICR according to RECIST v1.1
Disease Control Rate(DCR) | Up to 5 years
  Disease Control Rate(DCR) as Assessed by Investigator or BICR according to RECIST v1.1
Adverse Event | Up to 5 years
  Collect Serious Adverse Events (SAEs) and Adverse Events (AEs) from the time of signing the Informed Consent Form (ICF) until the safety follow-up visit.Evaluate the safety of the investigational drug.
Plasma Concentration of JS105 | Up to 3.5 years
  Collect JS105 PK sample to evaluate the blood drug concentration after the administration of JS105.

CONTACTS AND LOCATIONS:
Overall Officials: Xianming Luo, Doctor, Study Director — Medical Director
Locations (2):
- China (2):
  - Chinese Acadamy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - Henan Provincial Cancer Hospital, Zhengzhou, Henan